CLINICAL TRIAL: NCT03193463
Title: Pilot Trial of Intratumorally-Administered Topotecan Using Convection-Enhanced Delivery (CED) in Patients With Suspected Recurrent/Progressive World Health Organization (WHO) Grade III or IV (High Grade) Glioma Undergoing Stereotactic Biopsy (IND 117,240)
Brief Title: Intratumorally-Administered Topotecan Using CED in High Grade Glioma Undergoing Stereotactic Biopsy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Michael Vogelbaum, MD, PhD (Other)
Collaborators: Infuseon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Vogelbaum, MD, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INFT1317
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Glioma
Keywords: Topotecan; Convection-Enhanced Delivery
MeSH Terms: conditions — Glioma | interventions — Topotecan; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: There will be 3 arms to this study, and they will accrue independently of each other as they reflect distinctly separable populations of patients with rHGG.
  Arm 1: Predominantly enhancing mass with volume of 8 cc or less. Arm 2: Predominantly enhancing mass with volume of > 8 cc Arm 3: Predominantly non-enhancing mass
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Predominantly enhancing mass with volume of 8 cc or less (Experimental): Only 1 Cleveland Multiport Catheter (CMC) will be placed and CED will be performed intra-operatively only in a magnetic resonance imaging (MRI) equipped Operating Room. Topotecan infusion will be performed over a 4-hour period, with the goal of complete tumor coverage. The initial rate will be 1.20 ml/hour and infusion will be monitored by intermittent MRI imaging. The rate may be adjusted upwards during the infusion, in the event of incomplete tumor coverage, or downwards, if new mass effect is apparent. Following completion of the 4-hour infusion, the CMC will be removed. The initial rate for each subsequent patient may be adjusted upwards in increments of up to 1.20 ml/hour based upon the tumor coverage and safety characteristics of the previously treated patients.
  Interventions: Drug: Topotecan (<=8cc); Device: Cleveland Multiport Catheter; Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Predominantly enhancing mass with volume of > 8 cc (Experimental): 2 Cleveland Multiport Catheter (CMCs) will be placed and the total infusion rate of Topotecan per CMC to be used for the first 24 hours for the first patient will be 0.834 ml/hour (3.48 microliters/minute/microcatheter). The rate used for the second 24 hours of the infusion will be 1.668 ml/hour. If the first patient does not experience rate-limiting toxicity, then the patient #2's initial infusion rate will start at the highest tolerated rate for patient #1, and the second 24-hour rate for that patient will be increased by 0.834 ml/hour. Each subsequent patient will undergo rate escalation in a similar manner until we observe either: 1) complete coverage of the enhancing tumor by the infused Gadopentetic acid (Gd-DTPA), or 2) rate-limiting toxicity.
  Interventions: Drug: Topotecan (>8cc); Device: Cleveland Multiport Catheter; Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Predominantly non-enhancing mass (Experimental): The total infusion rate of Topotecan per Cleveland Multiport Catheter (CMC) to be used for the first 24 hours for the first patient will be 0.29 ml/hour. The rate used for the second 24 hours of the infusion will be 0.58 ml/hour. If the first patient does not experience rate-limiting toxicity, then the patient #2's initial infusion rate will start at the highest tolerated rate for patient #1, and the second 24-hour rate for that patient will be increased by 0.29 ml/hour. Each subsequent patient will undergo rate escalation in a similar manner until we observe either: 1) complete coverage of the non-enhancing tumor by the infused Gd-DTPA, or 2) rate-limiting toxicity.
  Interventions: Device: Cleveland Multiport Catheter; Diagnostic Test: Magnetic Resonance Imaging (MRI); Drug: Lower Does Topotecan

INTERVENTIONS:
Drug: Topotecan (<=8cc) — In predominantly enhancing mass with a volume of 8 cc or less of topotecan administered
  Other Names: Hycamtin
  Arms: Predominantly enhancing mass with volume of 8 cc or less
Drug: Topotecan (>8cc) — In predominantly enhancing mass with a volume of > 8 cc of topotecan administered. Initial rate is 0.834ml/hour with an increase to 1.668 ml/hour at the second infusion
  Other Names: Hycamtin
  Arms: Predominantly enhancing mass with volume of > 8 cc
Device: Cleveland Multiport Catheter — an investigational device, will be used to deliver the topotecan
Diagnostic Test: Magnetic Resonance Imaging (MRI) — to monitor the infusion of topotecan into the tumor
Drug: Lower Does Topotecan — Rate for non-enhancing tumors has an initial dose of 0.29ml/hour
  Other Names: Hycamtin
  Arms: Predominantly non-enhancing mass

SUMMARY:
The purpose of this study is to determine if treatment with topotecan by an alternative method, direct delivery into brain tumors, is safe and well tolerated. The Cleveland Multiport Catheter is a new, investigational device that will be used to deliver topotecan into your brain tumor. A second purpose of this study is to determine whether the Cleveland Multiport Catheter can be used effectively and safely to deliver topotecan into your brain tumor.

This study will also determine the best dose of topotecan to deliver to your tumor with use of the Cleveland Multiport Catheter and will also examine how your tumor responds to treatment with topotecan.

DETAILED DESCRIPTION:
Primary Objectives

* To investigate by MR imaging the spatial and temporal distribution of topotecan in enhancing or nonenhancing bulk tumor administered by convection-enhanced delivery (CED) in patients with recurrent/progressive WHO grade III or IV (high grade) glioma (HGG) who have failed standard therapy comprising surgical biopsy and/or resection and adjuvant chemotherapy and radiotherapy.
* To investigate by MR imaging the influence of the rate and topotecan concentration, on the spatial and temporal distribution of topotecan administered by CED in patients with with recurrent/progressive HGG

Secondary Objectives

* To investigate the extent to which backflow may be observed on MRI during CEDmediated delivery of topotecan
* To assess the safety, tolerability and toxicity profile of topotecan administered by CED using different doses and infusion rates.
* To observe evidence of activity of single-agent topotecan administered by CED to patients with recurrent/progressive HGG who have failed standard therapy comprising surgical biopsy and/or resection and adjuvant chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of supratentorial WHO Grade III or IV Glioma (High Grade Glioma) that has undergone surgical biopsy or resection followed by adjuvant chemoradiotherapy, that has evidence of recurrence or progression based on imaging studies and a stereotactic biopsy is indicated for confirmation of recurrence/progression
* Karnofsky Performance Status 70-100
* MRI demonstration of a stereotactically accessible enhancing mass that does not require resection to relieve clinically significant mass effect
* Patient understands the procedures and agrees to comply with the study requirements by providing written informed consent
* Laboratory values within the following ranges:

  * Absolute neutrophil count (ANC) ≥ 1,500 / μL
  * Platelet count ≥ 100,000 / μL
  * Hemoglobin ≥ 10 g / dL
  * prothrombin time (PT) / partial thromboplastin time (PTT) not above institutional norms
  * Estimated glomerular filtration rate (eGFR) of at least 50 mL/min

Exclusion Criteria:

* Patient is mentally or legally incapacitated at the time of the study
* Known HIV(+) or has been diagnosed with AIDS
* Participation in another investigational drug study in the prior 4 weeks
* Positive pregnancy test in a female
* Patient, in the opinion of the investigator, is likely to be poorly compliant
* Diffuse subependymal or cerebrospinal fluid (CSF) disease
* Tumors involving the cerebellum
* Tumor enhancement involving both hemispheres
* Active infection requiring treatment
* Unexplained febrile illness
* Radiation or chemotherapy within 4 weeks of enrollment
* Systemic diseases associated with unacceptable anesthesia or operative risk
* Inability to undergo magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Number of intra-operative catheter related complications | Up to 12 months
  Documentation of possible, probable, or definite catheter-related complications
Number of post-operative catheter related complications | Up to 12 months
  Documentation of possible, probable, or definite catheter-related complications
Number of catheter related complications after catheter removal | Up to 12 months
  Documentation of possible, probable, or definite catheter-related complications
Change in the spatial distribution of intratumorally-administered topotecan at serial timepoints using a gadolinium-based contrast agent, as determined by MRI scan | Up to 12 months
Changes in the spatial distribution of intratumorally-administered topotecan associated with changes in the infusion rate, as determined by MRI scan | Up to 12 months
Changes in the spatial distribution of intratumorally-administered topotecan at serial timepoints using volumetric magnetic resonance imaging, as determined by MRI scan | Up to 12 months
Changes in the spatial distribution of intratumorally-administered topotecan at serial timepoints using three-dimensional image reconstruction, as determined by MRI scan | Up to 12 months
Changes in the spatial distribution of intratumorally-administered topotecan associated with changes in the infusion concentration, as determined by MRI scan | Up to 12 months
Changes in the spatial distribution of intratumorally-administered topotecan associated with changes in the infusion duration, as determined by MRI scan | Up to 12 months

SECONDARY OUTCOMES:
Number of Participants with response as measured by the Response Assessment in Neuro-Oncology (RANO) Criteria | Up to 12 months
  Response includes objective response rate (ORR), median progression-free survival (PFS), proportion progression-free at six months (PFS-6), and median overall survival (OS)
Safety as measured by the common terminology criteria for adverse events (CTCAE) | Up to 12 months
  Safety will be determined through adverse events by arm

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Vogelbaum, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center